CLINICAL TRIAL: NCT07220733
Title: Safety and Feasibility of a Self-Balancing Exoskeleton for Rehabilitation in the Thoracic Surgical Intensive Care Unit: a Pilot Trial
Acronym: HEART
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP006
Record Dates: First submitted 2025-10-14; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Critical Illness; Post Operative Complication; Thoracic Surgery
Keywords: Thoracic Surgery; Postoperative Care; Atalante X Exoskeleton; Early Mobilisation; Intensive Care Unit (ICU)
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, unicentric, exploratory pilot study. All participants will receive the intervention (Atalante X exoskeleton sessions) in addition to standard ICU care. There is no randomization or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Early mobilization with the Atalante X self-balancing exoskeleton (Experimental): The Atalante X self-balancing exoskeleton is designed to support patients. The device enables patients to stand upright safely, to perform short steps (EarlyGait) or longer steps (RealGait), and to walk either in passive mode (with full assistance) or in active mode (with partial assistance depending on patient capacity). Sessions are delivered 2 to 3 times per week for up to 2 weeks or until ICU discharge. Each session starts with standing and progressively increases in intensity, with parameters such as duration, number of steps, verticalization time, and assistance level recorded. Training is conducted by certified staff, with the primary objective of evaluating safety and feasibility, and secondary outcomes including usability and preliminary effectiveness.
  Interventions: Device: Self-balancing robotic exoskeleton (Atalante X)

INTERVENTIONS:
Device: Self-balancing robotic exoskeleton (Atalante X) — This intervention consists of early mobilization sessions using the Atalante X, a self-balancing robotic exoskeleton (Wandercraft). Unlike other exoskeletons that require external support or crutches, this device is fully self-stabilizing and allows patients to stand and walk hands-free. It provides both passive and active modes, enabling short steps (EarlyGait) and longer steps (RealGait), with adjustable levels of assistance tailored to each patient's capacity. Sessions are performed 2-3 times per week for up to 2 weeks or until ICU discharge.

SUMMARY:
Patients admitted to the Intensive Care Unit (ICU) after thoracic surgery often experience complications related to immobility, such as muscle weakness, pulmonary issues, and longer recovery times. Early mobilization has been shown to improve outcomes, but its implementation is often limited by patient fragility and staff resources.

This study will test the safety and feasibility of using the Atalante X, a self-balancing exoskeleton, in the Thoracic Surgical ICU at Brigham and Women's Hospital. The exoskeleton is designed to support patients in standing and walking, even if they have limited strength or balance, thereby reducing the physical burden on healthcare staff and increasing patient mobility.

Eligible participants are adults recovering from thoracic surgery, who are debilitated (Johns Hopkins Highest Level of Mobility scale ≤ 5). Each participant will undergo up to 2-3 exoskeleton sessions per week for a maximum of 2 weeks. Sessions will be personalized, with progressive standing time and walking depending on patient tolerance.

The primary goal is to evaluate the safety of exoskeleton use, measured by adverse events such as skin lesions, cardiovascular instability, or accidental device-related issues.

The secondary goals are to evaluate:

Feasibility (ability to deliver sessions as planned, duration of standing/walking, level of assistance needed),

Usability (patient and staff satisfaction, ease of donning/doffing, staff workload), and

Preliminary effectiveness (improvement in mobility scores at discharge).

Results will provide early insights into whether robotic exoskeletons can be safely integrated into ICU rehabilitation programs after thoracic surgery.

DETAILED DESCRIPTION:
Prolonged bed rest and immobility are common in ICU patients and are strongly associated with poor outcomes, including pulmonary complications, neuromuscular weakness, cognitive impairment, and delayed recovery. Early mobilization after thoracic surgery has been demonstrated to improve respiratory function, reduce complications, and shorten hospital stays. However, significant barriers remain, including patient instability, staffing limitations, and the complexity of mobilizing critically ill patients with multiple devices and lines.

The Atalante X exoskeleton (Wandercraft, Paris, France) is a self-balancing robotic device that enables hands-free standing and walking. Using advanced AI-based algorithms, it adjusts to patient needs and provides variable assistance. Previous clinical studies in populations with spinal cord injury and post-stroke hemiplegia have shown the device to be safe and feasible, with improvements in mobility and balance. Atalante X has obtained FDA clearance (product code PHL, Class II, 21 CFR 890.3480).

This pilot study, named HEART (Hyper Early Atalante Rehabilitation Therapy), is a prospective, single-arm, unicentric exploratory trial conducted in the Thoracic Surgical ICU at Brigham and Women's Hospital (Boston, MA).

Expected impact:

This study will provide critical early data on the integration of robotic exoskeletons into ICU rehabilitation. By supporting patient mobilization earlier and more safely, Atalante X has the potential to improve outcomes after thoracic surgery, reduce ICU length of stay, and enhance patient recovery trajectories.

ELIGIBILITY:
Inclusion Criteria:

* Above age of 18 years old,
* Having undergone thoracic surgery that necessitated admission in the TSICU.
* Debilitated as defined as a JH-HLM score of 5 or less

Exclusion Criteria:

* Height < 6'3 feet or weight > 220 lbs restrictions
* Severe muscular spasticity of the lower extremities (Modified Ashworth Scale Grade 3 higher).
* Current fractures or incomplete bone junctions in the spine, pelvis, and/or lower extremities
* Osteoporosis or lower bone mineral density -3.5, and history(ies) of osteoporotic fracture(s).
* Skin disorders including Stage I pressure injuries at the hip, lower limbs, and Exoskeleton contact areas, according to the National and European Pressure Ulcer Classification System (NPUAP-EPUAP).
* Severe arthritis, acute arthritis, or synovitis after total or partial lower limb joint replacement.
* Myocardial infarction or angina or ischemic heart disease within the last 6 months.
* Uncorrectable leg length discrepancy over 2 cm when using additional correction tools.
* III-IV spine scoliotic deformity.
* Amputations and lower limb prostheses.
* Pregnancy
* Adults who lack the capacity to provide informed consent
* Cardiovascular instability as indicated by:
* Presence of unstable ventricular or atrial arrhythmias
* HR < 40 or HR > 140
* Lactate > 4.0 mmol/L
* On moderate-high dose vasopressors/inotropes
* Currently on VA ECMO
* Respiratory instability as indicated by:
* FiO2 > 0.6
* PEEP > 12 cm H2O
* RR > 35 bpm
* Currently on VV-ECMO
* Unable to follow commands
* Has bed rest orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of device- and procedure-related adverse events during exoskeleton use in ICU patients | Baseline and through study completion, an average of 2 weeks
  Safety will be assessed by the rate and type of device- and procedure-related adverse events during exoskeleton use. This includes skin lesions, catheter dislodgement, hemodynamic instability, falls, or any serious adverse events (SAEs or SADEs). An acceptable rate is defined as <15% overall and <15% for skin lesions.

SECONDARY OUTCOMES:
To evaluate the feasibility of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Compliance Measure Description: Compliance (%) = (number of completed exoskeleton sessions ÷ number of expected sessions) × 100. Expected sessions are fixed at 2 per week during the ICU stay. Sessions beyond 2 per week count as completed sessions but do not increase the expected total.
  Unit of Measure: percent (%)
To evaluate the feasibility of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Session Duration Measure Description: Duration of each exoskeleton session; mean duration per participant across all sessions.
  Unit of Measure: minutes
To evaluate the feasibility of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Total Steps per Session Measure Description: Number of steps completed during each exoskeleton session; mean steps per participant across sessions.
  Unit of Measure: steps
To evaluate the feasibility of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Duration by Walking Mode Measure Description: Time spent in each walking mode during exoskeleton sessions. EarlyGait and RealGait are reported separately; for each mode, the participant's mean duration across sessions is calculated.
  Unit of Measure: minutes
To evaluate the feasibility of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Steps by Walking Mode Measure Description: Number of steps performed in each walking mode during exoskeleton sessions. EarlyGait and RealGait are reported separately; for each mode, the participant's mean steps across sessions is calculated.
  Unit of Measure: steps
To evaluate the feasibility of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Lowest Assistance Level Achieved Measure Description: Lowest exoskeleton assistance (%) at which the participant completed ≥3 consecutive steps across all sessions.
  Unit of Measure: percent (%)
To evaluate the usability of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Donning and Doffing Time Measure Description: Time required to don and to doff the exoskeleton during each session. Donning and doffing are reported separately; for each, the participant's mean time across sessions is calculated.
  Unit of Measure: minutes
To evaluate the usability of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Satisfaction Score (Patient and Operator) Measure Description: Session-by-session satisfaction on a 0-10 numeric rating scale, reported by the patient and by the operator; mean per reporter (patient, operator) across sessions.
  Unit of Measure: score (0-10)
To evaluate the usability of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At study completion (average of 2 weeks)
  Outcome: Operator Workload (NASA-TLX) Measure Description: Overall workload scored with NASA-TLX at the end of the protocol.
  Unit of Measure: score (0-100)
To evaluate the usability of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At study completion (average of 2 weeks)
  Outcome: System Usability Scale (SUS) Measure Description: Device usability scored with the System Usability Scale at the end of the protocol.
  Unit of Measure: score (0-100)
To evaluate the usability of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | At each training session through study completion (average of 2 weeks)
  Outcome: Operators per Session (overall and by qualification) Measure Description: Total number of operators involved per session (donning, doffing, and during training). Counts will also be reported by qualification category (PT, RN, physician, technician, other). For each participant, the mean count per session will be calculated overall and per category.
  Unit of Measure: count and qualification
To evaluate the effectiveness of the self-balanced exoskeleton Atalante X among patients in the intensive care unit (ICU) who have undergone thoracic surgery | Baseline and at study completion (average of 2 weeks)
  Outcome: Functional Mobility (JH-HLM) Measure Description: Johns Hopkins Highest Level of Mobility score (1-8; higher = greater mobility), assessed per JH-HLM protocol.
  Unit of Measure: score (1-8)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States